CLINICAL TRIAL: NCT03467581
Title: Five-year Outcome of Laparoscopic Gastric Sleeve, Resolution of Comorbidities and Risk for Cumulative Nutritional Deficiencies.
Brief Title: Five-year Outcome of Laparoscopic Gastric Sleeve
Status: Recruiting | Type: Observational
Sponsor: Tartu University Hospital (Other)
Responsible Party: Principal Investigator, Eva-Maria Kikkas, Surgical resident, Tartu University Hospital
Other Study IDs: Sleeve5years
Record Dates: First submitted 2018-03-05; First posted 2018-03-16 (Actual); Last update posted 2018-03-16 (Actual); Status verified 2018-03

CONDITIONS: Bariatric Surgeries; Metabolic Surgery
Keywords: gastric sleeve

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to evaluate the long-term (5-year follow-up) results of laparoscopic gastric sleeve (LGS) in terms of weight loss and obesity related comorbidities, as well as the risk factors associated with postoperative nutritional deficiencies.

DETAILED DESCRIPTION:
The consecutive patients who undergo LGS for the treatment of morbid obesity at Tartu University Hospital are followed prospectively in cohort study. The outpatient hospital follow-up visits are conducted at 3 months, 1 year and 5 years postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* The criteria for bariatric surgery: BMI of >40, or >35 with certain obesity related comorbidities

Exclusion Criteria:

* Patients who did not fill the inclusion criteria

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who undergo LGS for the treatment of morbid obesity at Tartu University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2008-10-08 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Five-year outcome of laparoscopic gastric sleeve | 5-year follow-up
  5-year outcome in terms of weight loss, calculated in mean excess weight lost (%EWL).

SECONDARY OUTCOMES:
Five-year outcome of laparoscopic gastric sleeve | 5-year follow-up
  5-year outcome of resolution of obesity-related comorbidities (type 2 diabetes mellitus, hypertension, obstructive sleep apnea, dyslipidemia). Prevalence of comorbidities are presented in percentages. McNemar´s test is employed to analyse significance of resolution of comorbidities.
Five-year outcome of laparoscopic gastric sleeve | 5-year follow-up
  5-year risk for cumulative nutritional deficiencies. According to blood analysis results and patient provided information about taking supplementations (eg vitamine B12 or iron), prevalence of nutritional deficiencies are calculated in percetanges. Backward stepwise logistic regression is used to evaluate the risk factors for nutrition.

CONTACTS AND LOCATIONS:
Locations (1):
- Tartu University Hospital, Tartu, Estonia

IPD SHARING:
Plan to Share IPD: No